CLINICAL TRIAL: NCT01346839
Title: Effectiveness of Electronic Health Record-Based Interventions for Improving Follow-Up in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Scott and White Hospital & Clinic (Other)
Responsible Party: Principal Investigator, Hardeep, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-24978
Record Dates: First submitted 2011-02-23; First posted 2011-05-03 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Colon Cancer; Lung Cancer; Prostate Cancer
Keywords: Diagnostic delay; Prevention; Diagnostic errors
MeSH Terms: conditions — Colonic Neoplasms; Lung Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact Intervention (Experimental): The intervention will include activities such as electronic communication and surveillance that facilitate the care of patients experiencing delays. A trained chart reviewer will conduct chart reviews on trigger-positive patients to confirm they are at risk for care delays and this will be followed by an electronic and/or verbal communication to the provider. The intervention will be compared to usual care at both sites.
  Interventions: Behavioral: Contact Intervention
- Usual Care Control (No Intervention): The usual care at MEDVAMC consists of providers using an advanced EHR and its notification system (the View Alert system) that immediately alerts providers about clinically significant events. The system relies primarily on computerized notification (alerts) displayed prominently through a "View Alert" window that is displayed in the EHR every time a provider signs on or switches between patient records. The system does not require providers to read alerts, and providers do have an option of ignoring the View Alert window to bypass it. At SWHS there is a navigation program for patients who have received a cancer diagnosis by tissue biopsy. However, currently there is no routine tracking of patients if they do not show for their scheduled appointments and tests at SWHS.

INTERVENTIONS:
Behavioral: Contact Intervention — The intervention will include activities such as electronic communication and surveillance that facilitate the care of patients experiencing delays. A trained chart reviewer will conduct chart reviews on trigger-positive patients to confirm they are at risk for care delays and this will be followed by an electronic and/or verbal communication to the provider. The intervention will be compared to usual care at both sites.
  Arms: Contact Intervention

SUMMARY:
Diagnostic delays in ambulatory care are often due to breakdowns of related care processes. Electronic systems can improve follow-up and reduce delays by detecting missed appointments or incomplete procedures so that patients are called back to conduct timely investigations when appropriate. To achieve high standards of patient safety in cancer diagnosis, the investigators not only need to use information technology appropriately but also improve the processes, policies, and procedures of monitoring, communication, and coordination of care.

Given the importance of cancer-related diagnostic delays in ambulatory care, the investigators need effective methods to detect them, understand their causes, and intervene to reduce them. Manual techniques to detect these delays, such as spontaneous reporting and random chart reviews, have limited effectiveness. Our proposed study focuses on testing methods to proactively identify delays using certain "triggers" as they occur and intervene in a timely manner.

DETAILED DESCRIPTION:
The goal of this proposal is to demonstrate and test methods by which large health care systems can efficiently identify cancer patients who are more likely to experience diagnostic delays and pre-emptively rectify these delays. This study will build upon tools developed in our recent work (Aim1, prior IRB Protocol Number: H-23801) and test their effectiveness to identify patients at risk of experiencing delays in cancer diagnosis followed by an intervention that the investigators hypothesize will reduce these delays.

This is Aim 2 (for which the investigators are seeking approval) is the final Aim of this proposal. Aim 1 was approved under Protocol Number: H-23801.

In Aim 2 the investigators will determine the effectiveness of an IT-based intervention (consisting of data mining using triggers tested in Aim 1 followed by targeted electronic communication and surveillance techniques) to facilitate cancer diagnosis as compared with usual care (no use of trigger or electronic communication and surveillance). Hypothesis 1: The time from first appearance of a diagnostic clue to follow-up action (e.g. colonoscopy performance after a positive FOBT) will be significantly less in the intervention arm than in usual care. Hypothesis 2: The percentage of patients receiving timely follow-up care will be significantly more in the intervention arm than in usual care. To improve the generalizability of our findings to multiple ambulatory care environments, the investigators will conduct our research in two settings: an urban Veterans Affairs facility in Houston, Texas and a large primary care network in central Texas. These settings include internal medicine and family medicine, academic and nonacademic practices, and significant racial, gender, ethnic, age, urban/rural, and socioeconomic diversity. Our study addresses coordination and timeliness of care, both of which are priorities to achieve high quality care.

Hypothesis 3: Overall, the trigger will achieve a positive predictive value (PPV) of at least 50% in identifying delays in care. PPV is defined as the number of charts correctly identified with a delay in diagnostic evaluation, divided by the total number of charts identified by the trigger, and was deemed to be the approximately level necessary to avoid substantial contribution to provider alert fatigue.

ELIGIBILITY:
Inclusion Criteria:

All primary care providers at both study sites who agree to be in the study. Intervention will be performed on those whose patients are electronically identified to have suspected cancer defined as presence of any predefined clue for cancer that is not followed-up in a timely manner. Three cancers are included; colorectal, lung and prostate and their clues include • chest x-imaging suspicious for malignancy • suspected or confirmed iron deficiency anemia • positive FOBT • hematochezia • abnormal PSA Patients will be selected from the data warehouse .

Exclusion Criteria:

Primary care providers who do not wish to be in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1256 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hardeep Singh, MD MPH, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas

REFERENCES:
- [Derived] Murphy DR, Wu L, Thomas EJ, Forjuoh SN, Meyer AN, Singh H. Electronic Trigger-Based Intervention to Reduce Delays in Diagnostic Evaluation for Cancer: A Cluster Randomized Controlled Trial. J Clin Oncol. 2015 Nov 1;33(31):3560-7. doi: 10.1200/JCO.2015.61.1301. Epub 2015 Aug 24. PMID 26304875

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contact Intervention | Usual Care Control
Started | 683 | 573
Completed | 369 | 364 (All triggers were applied retrospectively on 7/19/2012.)
Not Completed | 314 | 209

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contact Intervention | Usual Care Control | Total
Number analyzed (Participants) | 369 | 364 | 733
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (7.4) | 60.3 (8.5) | 60.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 66 | 104
  Male | 331 | 298 | 629
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 33 | 68
  Not Hispanic or Latino | 334 | 331 | 665
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 13 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 141 | 154 | 295
  White | 213 | 179 | 392
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 17 | 27
Region of Enrollment [Number; unit: participants]
  United States | 369 | 364 | 733
Number of Comorbidities [Mean (Standard Deviation); unit: Comorbidities] | 2.2 (1.3) | 2.1 (1.4) | 2.2 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Differences in Time to Documented Follow-up of a Red Flag Suggestive of Cancer
Description: Differences between the intervention and control groups (based on a Cox Proportional Hazards Survival Analysis) in median time to documented follow-up of a red flag (e.g., colonoscopy performance after positive FOBT) or of a deliberate decision by the treating provider not to take follow-up action. When less than 50% of patients in either group received diagnostic evaluation (ie, medians were not reached), the point at which 40% received diagnostic evaluation was compared instead.
Time Frame: 15 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Contact Intervention | Usual Care Control
Number analyzed (Participants) | 369 | 364
Days
  Time to Follow-up of Colorectal Trigger | 104 [91.2 to 116.8] | 200 [162.5 to 210.0]
  Time to Follow-up of Prostate Trigger | 144 [131.2 to 153.1] | 192 [182.0 to 199.1]
  Time to Follow-up of Lung Trigger | 65 [50.4 to 79.6] | 93 [70.3 to 115.7]
Statistical Analysis 1: Comparison: Contact Intervention vs Usual Care Control; Test type: Superiority or Other; p < 0.05, Regression, Cox

2. Secondary Outcome: Percentage of Patients Receiving Timely Follow-up of a Red Flag Suggestive of Cancer
Description: The percentage of patients receiving timely follow-up care, as defined by action taken by provider within appropriate pre-defined time intervals for each diagnostic clue, in both intervention and control groups.
Time Frame: 15 months
Measure: Number; unit: percentage of follow-up
Arm/Group | Contact Intervention | Usual Care Control
Number analyzed (Participants) | 369 | 364
percentage of follow-up | 73.4 | 52.2

3. Secondary Outcome: Percentage of Cases With no Documented Justification for no Follow-up
Description: This is a descriptive sub-analysis looking only at cases with no follow-up at the end of the follow-up period. Specifically, out of the cases that never got follow-up, this represents the percent of that subsample that had no justification in the medical record for the lack of follow-up. This is based on manual chart reviews.
Time Frame: 15 months
Measure: Number; unit: percentage with no documentation
Arm/Group | Contact Intervention | Usual Care Control
Number analyzed (Participants) | 174 | 98
percentage with no documentation | 33.9 | 48.0

4. Secondary Outcome: Number of Participants Diagnosed With Cancer After Delay in Diagnostic Evaluation
Description: Subsequent diagnosis of nonmalignant neoplasia, cancer, or death, and treatments required as a result of new cancer diagnoses after a pre-specified interval.
Time Frame: 15 months
Measure: Number; unit: Number of patients diagnosed with cancer
Arm/Group | Contact Intervention | Usual Care Control
Number analyzed (Participants) | 369 | 364
Number of patients diagnosed with cancer | 13 | 10

5. Secondary Outcome: Trigger Positive Predictive Value
Description: Positive Predictive Values of each of the triggers in identifying patients with a true delay in diagnostic evaluation. Calculated as: percentage of patients identified as trigger positive that actually had a delay.
Time Frame: 15 months
Measure: Number; unit: Percentage of participants
Arm/Group | Contact Intervention | Usual Care Control
Number analyzed (Participants) | 369 | 364
Percentage of participants | 63.5 | 55.3

ADVERSE EVENTS:
Arm/Group | Contact Intervention | Usual Care Control
Serious Adverse Events (participants affected / at risk) | 0/369 | 0/364
Other Adverse Events (participants affected / at risk) | 0/369 | 0/364

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No